CLINICAL TRIAL: NCT01315067
Title: Non-invasive Diagnosis of Acute Rejection in Renal Transplant Patients Using Mass Spectrometry of Urine Samples - a Multicentre Diagnostic Phase III Trial
Brief Title: Diagnosis of Acute Rejection in Renal Transplant Patients by Urine Mass Spectrometry
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Wilfried Gwinner, Prof. Dr. med., Hannover Medical School
Other Study IDs: MS-GW4/6-1
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Rejection of Renal Transplant
Keywords: kidney transplantation; acute rejection; diagnosis; urine analysis; urinary peptides; mass spectrometry; allograft biopsy; pathology; diagnostic study
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine samples, kidney allograft biopsies
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Reliable and timely detection of acute rejections in renal transplant patients is important to preserve the graft function and to prevent premature graft failure. The current gold standard for the rejection diagnosis is a renal biopsy which is usually performed upon an unexplained decline in the graft function (determined by serum creatinine or clearance). Because of the insensitivity of creatinine determinations and the invasiveness of renal biopsies, non-invasive tests have been suggested to diagnose acute rejection including mass spectrometry (MS) analysis of urine samples.

The ability of MS analysis to detect acute rejection has been demonstrated in small studies on selected patients but evidence is lacking that this test is efficacious in the routine setting of the post-transplant patient care. Based on our previous work that established urine peptide sets for acute rejection by MS, a prospective, multicentre diagnostic phase III study will be executed.

The aim of the study is to prove that this test is as equally effective as the allograft biopsy to detect acute rejection in patients that undergo a biopsy for unexplained renal dysfunction. The perspective of this approach is that the test could be used either in place of the biopsy or as decision guidance whether a biopsy is necessary to confirm the presence of rejection. Another perspective is that the MS test (respectively, a simplified test system derived from this method) could be used in the regular post-transplant surveillance for acute rejection, in place of the relatively insensitive procedure with periodic monitoring of the graft function by creatinine determinations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a kidney or combined kidney/pancreas transplantation
* Unexplained renal allograft dysfunction within the first year of transplantation
* Renal allograft biopsy, which is clinically indicated to verify or exclude an acute rejection

Exclusion Criteria:

* Lacking consent of the patient to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a kidney or combined kidney/pancreas transplantation from several German transplant centres with an acute unexplained allograft dysfunction within the first year of transplantation who require a clinically indicated allograft biopsy
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2011-10; Primary Completion 2017-03 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Ability of the urine mass spectrometry test to diagnose acute renal allograft rejection, compared to the gold standard 'allograft biopsy' | Results of the urine test will be assessed in relation to the simultaneously performed allograft biopsy (1 day)
  In patients with unexplained renal allograft dysfunction who get an allograft biopsy to clarify if an acute rejection is present, a simultaneous urine sample will be taken.
  The peptide pattern of this urine sample is analyzed by mass spectrometry and a diagnosis is made (rejection present/not present) based on a pre-defined peptide pattern which was established to detect acute allograft rejection.
  In the primary outcome analysis, the sensitivity and specificity of the rejection diagnosis by the urine test is compared to the diagnosis made by the allograft biopsy.

SECONDARY OUTCOMES:
Sensitivity and specificity of the urine test to diagnose acute renal allograft rejection in subgroups with different severity grades of the rejection | Results of the urine test will be assessed in relation to the simultaneously performed allograft biopsy (1 day)
  Sensitivity/specificity measures for the urine test will be determined in subgroups of patients with different severity of the rejection. Severity grading is based on the pathomorphological classification of the rejection (according to the BANFF classification) and on the functional impairment of the allograft at the time of rejection diagnosis.
Sensitivity and specificity of the urine test to diagnose acute renal allograft rejection in subgroups with kidney transplantation alone and with combined pancreas/kidney transplantation | Results of the urine test will be assessed in relation to the simultaneously performed allograft biopsy (1 day)
  Sensitivity/specificity measures for the urine test will be determined in subgroups of patients who have a kidney transplant or a combined pancreas/kidney transplant.
Sensitivity and specificity of the urine test to diagnose acute renal allograft rejection in subgroups with concurrent infection | Results of the urine test will be assessed in relation to the simultaneously performed allograft biopsy (1 day)
  Sensitivity/specificity measures for the urine test will be determined in subgroups of patients who have concurrent infections at the time of the biopsy and urine sampling such as cytomegaly virus, polyoma virus, and urinary tract infection. The analysis intends to identify potential interference of these conditions with the urine mass spectrometry test.

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Gwinner, Prof. /MD, Principal Investigator — Hannover Medical School
Locations (8):
- Germany (8):
  - RTW University of Aachen, Aachen
  - Charite Universitätsmedizin Berlin, Berlin
  - Kliniken der Stadt Köln gGmbH, Cologne
  - University of Erlangen-Nuremberg, Erlangen
  - Universitätsklinikum Essen, Essen
  - Hannover Medical School, Hanover
  - Universitätsklinikum Jena, Jena
  - Ludwig-Maximilians-Universitätsklinik München, München

REFERENCES:
- [Background] Wittke S, Haubitz M, Walden M, Rohde F, Schwarz A, Mengel M, Mischak H, Haller H, Gwinner W. Detection of acute tubulointerstitial rejection by proteomic analysis of urinary samples in renal transplant recipients. Am J Transplant. 2005 Oct;5(10):2479-88. doi: 10.1111/j.1600-6143.2005.01053.x. PMID 16162198
- [Background] Metzger J, Chatzikyrkou C, Broecker V, Schiffer E, Jaensch L, Iphoefer A, Mengel M, Mullen W, Mischak H, Haller H, Gwinner W. Diagnosis of subclinical and clinical acute T-cell-mediated rejection in renal transplant patients by urinary proteome analysis. Proteomics Clin Appl. 2011 Jun;5(5-6):322-33. doi: 10.1002/prca.201000153. Epub 2011 Apr 29. PMID 21538920
- [Derived] Zapf A, Gwinner W, Karch A, Metzger J, Haller H, Koch A. Non-invasive diagnosis of acute rejection in renal transplant patients using mass spectrometry of urine samples - a multicentre phase 3 diagnostic accuracy study. BMC Nephrol. 2015 Sep 15;16:153. doi: 10.1186/s12882-015-0146-x. PMID 26374548